CLINICAL TRIAL: NCT03368651
Title: The Impact on Survival of Neo-adjuvant Transarterial Chemoinfusion (TAI) for Patients With Hepatocellular Carcinoma And Portal Vein Tumor Thrombosis (PVTT) Who Underwent Hepatectomy : A Random, Controlled, Stage III Clinical Trial.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rong-ping Guo, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2017-076-01
Record Dates: First submitted 2017-12-04; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): transarterial chemoinfusion (TAI) with mFOLFOX6 (oxaliplatin, calcium folinate, and 5-FU)
  Interventions: Procedure: TAI
- control group (No Intervention): no neo-adjuvant treatment before operation

INTERVENTIONS:
Procedure: TAI — transarterial chemoinfusion with mFOLFOX6 (oxaliplatin, calcium folinate, and 5-FU)
  Arms: treatment group

SUMMARY:
To compare the impact on survival of neo-adjuvant TAI for patients with HCC and PVTT who underwent hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old and younger than 75 years;
* ECOG PS≤1;
* proven hepatocellular carcinoma according patological examination or EASL/AASLD diagnostic criteria;
* not previous treated for tumor;
* estimated tumor and tumor thrombosis could be removed en bloc in operation;
* no distant metastasis;
* the lab test could meet: neutrophil count≥2.0×109/L; hemoglobin≥100g/L; platelet count≥75×109/L; serum albumin≥35g/L; total bilirubin<2-times upper limit of normal; ALT<3-times upper limit of normal; AST<3-times upper limit of normal; serum creatine<1.5-times upper limit of normal; PT≤upper limit of normal plus 4 seconds; INR≤2.2;
* sign up consent;

Exclusion Criteria:

* cannot tolerate TAI or surgery;
* distant metastasis exits;
* known history of other malignancy;
* be allergic to related drugs;
* underwent organ transplantation before;
* be treated before (interferon included);
* known history of HIV infection;
* known history of drug or alcohol abuse;
* have GI hemorrhage or cardiac/brain vascular events within 30 days;
* pregnancy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 60 months
  overall survival

SECONDARY OUTCOMES:
recurrence-free survival (RFS) | From date of randomization until the date of recurrence, assessed up to 60 months
  recurrence-free survival
recurrence rate | 1 year, 2 year, 3 year, 5 year after surgery
  recurrence rate

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided